CLINICAL TRIAL: NCT05074095
Title: Injuries of the Urogenital Tract in Polytraumatized Patients in Correlation With Injuries to the Spine and Pelvic Girdle- Are There Positive Predictive Factors
Brief Title: Analysis of Urogenital Injuries in Polytraumatized Patients
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: 229/20 S-EB
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Polytrauma
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Patients with urogenital injuries
  Interventions: Other: retrospective analysis
- 2: Patients without urogenital injuries
  Interventions: Other: retrospective analysis

INTERVENTIONS:
Other: retrospective analysis

SUMMARY:
Urogenital injuries occur in approximately 5-10 % of all severly injured patients. The literature lacks a thorough investigation into the mechanisms of trauma, the analysis of the whole urogenital tract and especially the correlation of thoracic and lumbar spine and pelvic injuries with urogenital injuries.

The goal of this study is to provide a thorough investigation into these primary end points in a multicenter study of university hospitals in Germany.

ELIGIBILITY:
Inclusion Criteria:

* ISS (Injury severity score) > 15 points
* Patient Age > 16
* Fracture of the thoracic and/ or lumbar spine
* Fracture of the pelvic girdle
* at least one AIS (abbreviated injury scale) > 2

Exclusion Criteria:

* ISS < 16 points
* no fractures of the thoracic or lumbar spine or fractures of the pelvic girdle
* no AIS > 2
* patient age under 16 years of age

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective analysis of polytrauma patients.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Predictive factors for urogenital injuries | 5 years
  This retrospective analysis is designed to identify predictors of urogenital injuries in polytrauma patients

IPD SHARING:
Plan to Share IPD: No